CLINICAL TRIAL: NCT03097393
Title: Serum Procalcitonin Level May Predict Acute Kidney Injury in ICU Patients With Sepsis
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Mahmoud Hamada imam, Lecturer in Internal Medidicne Department- Faculty of Medicine, Benha University
Other Study IDs: Benha317
Record Dates: First submitted 2017-03-25; First posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AKI GROUP: measure Procalcitonin among Patient developed Acute kidney injury during ICU stay
  Interventions: Diagnostic Test: measure Serum procalcitonin level
- Non-AKI group: measure Procalcitonin among Patient did not develop Acute kidney injury during ICU stay
  Interventions: Diagnostic Test: measure Serum procalcitonin level

INTERVENTIONS:
Diagnostic Test: measure Serum procalcitonin level — measuring procalcitonin level

SUMMARY:
The aim of this study is to examine if procalcitonin (PCT) can be used for early prediction of AKI septic patients in ICU.

DETAILED DESCRIPTION:
67 patients with sepsis were enrolled in this study. On admission, PCT was measured together with serum creatinine, urea, and other inflammatory markers. Quick Sepsis-related Organ Failure Assessment was calculated at the emergency department. Patients were classified into those with Acute kidney injury (AKI) and non-AKI groups.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients with sepsis

Exclusion Criteria:

* Patient known to have End-stage kidney disease
* Patients on Renal replacement therapy
* patients without procalcitonin level within 24 hours from admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients with sepsis
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
development of AKI | 28 Days
  elevated kidney functions creatinine or oliguria

IPD SHARING:
Plan to Share IPD: No